CLINICAL TRIAL: NCT02770911
Title: Anastomotic Leakage in Laparoscopic Anterior Resection With or Without "Dog Ear" Double-stapled Anastomosis for Rectal Cancer : A Prospective, Randomized, Controlled Study
Brief Title: Laparoscopic Anterior Resection With or Without "Dog Ear" Double-stapled Anastomosis for Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Guoxian Guan, Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJMU-20160424
Record Dates: First submitted 2016-05-08; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Rectal Carcinoma; Laparoscopy; Anastomotic Leak
Keywords: Rectal Carcinoma; Laparoscopy; Anastomotic Leak; Double-stapling technique
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without "Dog Ear" group (Experimental): Before anastomosis, the surgeon made a laparoscopic suturing on the two dog ears by using 3-0 monofilament sutures, and pull two dogears of staple line around the trocar by a tied suture through two dog ears. By this way, the staple line was kept within the circular knife when the circular stapler was closed. Then a true end-to-end anastomosis was performed after stapler firing.
  Interventions: Procedure: without "Dog Ear" group
- with "Dog Ear" group (Active Comparator): traditional double-stapled anastomosis was used for laparoscopic anterior resection
  Interventions: Procedure: with "Dog Ear" group

INTERVENTIONS:
Procedure: without "Dog Ear" group — a modified double-stapling technique with eliminating the dogears in laparoscopic anterior resection
  Other Names: modified laparoscopic double-stapled anastomosis
  Arms: without "Dog Ear" group
Procedure: with "Dog Ear" group — a traditional double-stapling technique without eliminating the dogears in laparoscopic anterior resection
  Other Names: traditional laparoscopic double-stapled anastomosis
  Arms: with "Dog Ear" group

SUMMARY:
The study evaluates the feasibility and advantage of modified laparoscopic double-staple anastomosis technique which to eliminate the 'dog ears' in laparoscopic rectal anterior resection.

DETAILED DESCRIPTION:
Laparoscopic surgeons commonly make rectal transection intracorporeally by laparoscopic linear stapler during rectal anterior resection and perform an end-to-end anastomosis by circular stapler. But the so-called 'dog ears', two stapled corners of the rectal stump after laparoscopic linear transection of rectum, are very common. The lateral intersections of double-stapled anastomoses are structural weak spot area, and they are considered to be the potential ischemic areas leading to anastomosis leakage and the possible sites occurring local recurrence. Previous study reported a modified technique for rectal reconstruction during open surgery, and they could use circular stapler to eliminate the staple line on the rectal stump and cut off the 'dog ears'. But because of the narrow pelvic cavity, it is very difficult to perform this technique in laparoscopic rectal surgery and there is no related report on laparoscopic application. In this study, we evaluates the feasibility and advantage of modified laparoscopic double-staple anastomosis technique, to eliminate the "dog ears" in laparoscopic rectal anterior resection by laparoscopic suturing on the staple line.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility rule of enrollment
* Rectal adenocarcinoma above the peritoneal reflection
* at least 18 years old & at most 80 years old
* Clinically diagnosed cT1-T4aN0-2 disease
* no contraindication to laparoscopic surgery
* without other malignancies in medical history

Exclusion Criteria:

* concurrent or previous diagnosis of invasive cancer within 5 years
* locally advanced cancers requiring en bloc multivisceral resection
* intestinal obstruction
* intestinal perforation
* American Society of Anesthesiologists(ASA) class 4 or 5
* pregnant or breast-feeding women
* history of mental disorder
* participation in another rectal cancer clinical trial relating to surgical technique

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
anastomotic leakage rate | 30 days since the date of surgery

SECONDARY OUTCOMES:
Intra-operative and post-operative complications | 30 days since the date of surgery
post-operative Mortality | 30 days since the date of surgery
re-operation rate | 30 days since the date of surgery
QLQ 30 | at postoperative 3,6 and 12 months
Wexner's scoring | at postoperative 3,6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guo-xian Guan, MD,PhD, Principal Investigator — Fujian Medical University Union Hospital

REFERENCES:
- [Result] Roumen RM, Rahusen FT, Wijnen MH, Croiset van Uchelen FA. "Dog ear" formation after double-stapled low anterior resection as a risk factor for anastomotic disruption. Dis Colon Rectum. 2000 Apr;43(4):522-5. doi: 10.1007/BF02237198. PMID 10789750
- [Result] Kang J, Lee HB, Cha JH, Hur H, Min BS, Baik SH, Kim NK, Sohn SK, Lee KY. Feasibility and impact on surgical outcomes of modified double-stapling technique for patients undergoing laparoscopic anterior resection. J Gastrointest Surg. 2013 Apr;17(4):771-5. doi: 10.1007/s11605-012-2122-0. Epub 2013 Jan 4. PMID 23288715
- [Result] Kim HJ, Choi GS, Park JS, Park SY. Comparison of intracorporeal single-stapled and double-stapled anastomosis in laparoscopic low anterior resection for rectal cancer: a case-control study. Int J Colorectal Dis. 2013 Jan;28(1):149-56. doi: 10.1007/s00384-012-1582-8. Epub 2012 Sep 27. PMID 23014975
- [Result] Chen ZF, Liu X, Jiang WZ, Guan GX. Laparoscopic double-stapled colorectal anastomosis without "dog-ears". Tech Coloproctol. 2016 Apr;20(4):243-7. doi: 10.1007/s10151-016-1437-3. Epub 2016 Feb 22. No abstract available. PMID 26902367
- [Result] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450